CLINICAL TRIAL: NCT05366192
Title: The Safety of Paxlovid (Nirmatrelvir/Ritonavir) in Hemodialysis Patients With SARS-CoV-2 Infection
Brief Title: The Safety of Paxlovid in Hemodialysis Patients With Covid-19
Acronym: SPHPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-0067
Record Dates: First submitted 2022-04-28; First posted 2022-05-09 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Safety Issues
MeSH Terms: interventions — nirmatrelvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Paxlovid stage 1 group (Experimental): Subjects in stage 1 will be treated with nirmatrelvir 150mg qd (another 75mg will be supplied after hemodialysis treatment) and ritonavir 100mg bid everyday for 5 days.
  Interventions: Drug: Nirmatrelvir and ritonavir stage 1
- Paxlovid stage 2 group (Experimental): In stage 2, subjects will be treated with nirmatrelvir 300mg qd (another 150mg will be supplied after hemodialysis treatment) and ritonavir 100 bid everyday for 5 days.
  Interventions: Drug: Nirmatrelvir and ritonavir stage 2

INTERVENTIONS:
Drug: Nirmatrelvir and ritonavir stage 1 — Nirmatrelvir 150mg qd (another 75mg will be supplied after hemodialysis treatment) and ritonavir 100mg bid everyday for 5 days.
  Other Names: small dose
  Arms: Paxlovid stage 1 group
Drug: Nirmatrelvir and ritonavir stage 2 — Nirmatrelvir 300mg qd (another 150mg will be supplied after hemodialysis treatment) and ritonavir 100 bid everyday for 5 days.
  Other Names: high dose
  Arms: Paxlovid stage 2 group

SUMMARY:
Infection with SARS-CoV-2 continue to threaten global health. Persons with chronic kidney disease, including dialysis treatment are at hight risk for severe Covid-19 and associated adverse outcomes. Paxlovid (Nirmatrelvir/Ritonavir) decreases risk of progression to severe Covid-19. It is not recommended for dialysis patients because due to lack of data. The aim of the present study is evaluate the safety of Paxlovid in hemodialysis patients with SARS-CoV-2 infection.

This is a prospective study. In stage 1 arm, 10 hemodialysis patients with SARS-COV-2 infection will be treated with nirmatrelvir 150mg qd (another 75mg will be supplied after hemodialysis treatment) and ritonavir 100mg bid everyday for 5 days. In stage 2 arm, 10 patients will be treated with nirmatrelvir 300mg qd (another 150mg will be supplied after hemodialysis treatment) and ritonavir 100 bid everyday for 5 days. The primary outcome is the number of patients whose ALT, AST or total bilirubin increase two times from baseline. The secondary outcome is the number of patients whose SARS-CoV-2 lower than 500 copies/mL.

DETAILED DESCRIPTION:
This is a prospective, two arms (two stage) study. There will be include 20 subjects. The including criteria are 1.Understand the present study/Agree and sign informed consent; 2. Age is between 18 and 75 men or women at the screening; 3.Blood purification twice or three times/week, including hemodialysis, hemofiltration, hemodiafiltration, CRRT or hybrid blood purification; 4.Regular hemodialysis≥1 month; 5.Patients with arteriovenous fistula or artificial arteriovenous fistula; 6. Patients infected with SARS-CoV-2 and the CT value of nucleic acid detection<35. The exclusion criteria are 1.Blood purification treatment<1month; 2.Liver function (ALT or AST) is three times the upper the normal; 3.The severe or critical patients with Covid-19; 4.Patients who are treated with medicines that highly dependent on CYP3A, including but not limit to afzosin, pethidine, ranolazine, amiodarone, propafenone, quinidine, fusidic acid, voriconazole, terfenadine, colchicine, rifabutin, clozapine, dihydroergot, cisapride, simvastatin, diazepam, salbutam, triazolam, carbamazepine, phenobarbital, rifampicin; 5.Patients with galactose intolerance; 6. Pregnant and lactating women; 7.Patients was allergic to paxlovid; 8.Participating in other intervention studies; 9.The investigator judged that the condition of the subjects was not suitable for the study.

Subjects in stage 1 arm will be treated with nirmatrelvir 150mg qd (another 75mg will be supplied after hemodialysis treatment) and ritonavir 100mg bid everyday for 5 days. In stage 2 arm subjects will be treated with nirmatrelvir 300mg qd (another 150mg will be supplied after hemodialysis treatment) and ritonavir 100 bid everyday for 5 days. All of subjects will received hemodialysis two times during the study.

The primary outcome is the number of patients whose ALT, AST or total bilirubin increase two times from baseline. The secondary outcome is the number of patients whose SARS-CoV-2 lower than 500 copies/mL.

ELIGIBILITY:
Inclusion Criteria:

* 1.Understand the present study/Agree and sign informed consent.
* 2.Age is between 18 and 75 at the screening
* 3.Blood purification twice or three times/week, including hemodialysis, hemofiltration, hemodiafiltration, CRRT or hybrid blood purification.
* 4.Regular hemodialysis≥1 month
* 5.Patients with arteriovenous fistula or artificial arteriovenous fistula.
* 6.Patients infected with Covid-19, the PCR CT value of nucleic acid detection<35.

Exclusion Criteria:

* 1.Blood purification treatment<1month.
* 2.Liver function (ALT or AST) is three times the upper the normal.
* 3.The severe or critical patients with Covid-19.
* 4.Drug that highly dependent on CYP3A, including but not limit to afzosin, pethidine, ranolazine, amiodarone, propafenone, quinidine, fusidic acid, voriconazole, terfenadine, colchicine, rifabutin, clozapine, dihydroergot, cisapride, simvastatin, diazepam, salbutam, triazolam, carbamazepine, phenobarbital, rifampicin.
* 5.Patients with galactose intolerance.
* 6. Pregnant and lactating women.
* 7.Patients was allergic to paxlovid.
* 8.Participating in other intervention studies.
* 9.The investigator judged that the condition of the subjects was not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Change of Liver function | 5 days
  Number of patients whose ALT, AST or total bilirubin increase 2 times from baseline

SECONDARY OUTCOMES:
The effectiveness of Paxlovid | 5 days
  Number of patients whose SARS-CoV-2 lower than 500copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Leyi Gu, Principal Investigator — Renal Division, Renji Hospital
Locations (1):
- Department of Nephrology, Renji Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
When the study is complete, the clinical study report will be shared.
Supporting Information: CSR
Time Frame: September, 2022
Access Criteria: Publication